CLINICAL TRIAL: NCT04144699
Title: Clinical Validation of Omron WheezeScan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Omron Healthcare Co., Ltd. (Industry)
Collaborators: University of Wisconsin, Madison (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: HDV-CDD-190046
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Asthma in Children; Bronchitis; Bronchiolitis
Keywords: wheeze; rhonchus
MeSH Terms: conditions — Bronchitis; Bronchiolitis; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Wheezing 3~11months: Patient has wheezing, age 3 to 11 months
- Wheezing 12~23months: Patient has wheezing, age 12 to 23 months
- Wheezing 24~35months: Patient has wheezing, age 24 to 35 months
- Wheezing 36~107months: Patient has wheezing, age 36 to 107 months
- No wheezing 3~11months: Patient do not have wheezing, age 3 to 11 months
- No wheezing 12~23months: Patient do not have wheezing, age 12 to 23 months
- No wheezing 24~35months: Patient do not have wheezing, age 24 to 35 months
- No wheezing 36~107months: Patient do not have wheezing, age 36 to 107 months

SUMMARY:
The WheezeScan sensitivity and specificity are set to statistically prove equal to or higher values than the predicate PulmoTrack device model 2020.

ELIGIBILITY:
Inclusion Criteria:

Mild to moderate diagnosed or suspected asthma, bronchitis, or bronchiolitis patients who meet all of the following criteria are considered as eligible.

1. Does the subject have mild to moderate diagnosed or suspected asthma, bronchitis, or bronchiolitis?
2. Is the subject between the ages of 3 months to 8 years old?
3. Is the parent or legal guardian available, and capable and willing to give a consent on the child's behalf.

Exclusion Criteria:

The subjects will be excluded from the study, if they have any of the following criteria.

1. Does the subject have skin rashes or wounds on the chest?
2. Does the subject have known allergies or irritant contact dermatitis or having hypersensitive skin?
3. Does the subject have a defibrillator and/or pacemaker (which could interfere with the sounds to be detected)?
4. Does the subject have an allergy to disinfecting alcohol?
5. Does the subject have wheezes caused by not asthma, such as reflux esophagitis, pneumonia, vocal cord dysfunction, Tracheomatosis?
6. Does the subject have a heavy runny nose?
7. Is it difficult to hear auscultation due to the subject fussing, crying or vocalizing at data collection?
8. Is the subject having difficulty breathing or having severe symptoms?
9. Was the subject enrolled more than once for the same resulted breath sounds?

   * Note: The subject maybe enrolled once per arm (once wheezing, once non-wheezing).

Ages: 3 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Wheezing Total : Min.120, Wheezing 3~11months : Min.19, Wheezing 12~23months : Min.19, Wheezing 24~35months : Min.19, Wheezing 36~107months : Min.38, No wheezing total : Min.120, No wheezing 3~11months : Min.19, No wheezing 12~23months : Min.19, No wheezing 24~35months : Min.19, No wheezing 36~107months : Min.38
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the sensitivity and specificity of the Omron WheezeScan device | Novemver 1, 2019 ~ November 30, 2021
  The WheezeScan device will be compared to the gold standard, auscultation, which will be performed by a physician or a qualified healthcare professional with a minimum of 3 years' experience. All breath sounds will be recorded for comparison in case of discrepancy.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Tekton Research, Chamblee, Georgia
  - University of Chicago, Chicago, Illinois
  - PMG Research of DuPage, Joliet, Illinois
  - Long Island Jewish Medical Center, New York, New York
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - PMG Research of Charleston, Charleston, South Carolina
  - Meridian Clinical Research, LLC, Dakota Dunes, South Dakota
  - PMG Research of Bristol, Bristol, Tennessee
  - PMG Research of Knoxville, Jefferson City, Tennessee
  - Tekton Research, Beaumont, Texas
  - Tekton Research, San Antonio, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No plan to share the data